CLINICAL TRIAL: NCT00370396
Title: To Assess the Safety, Reactogenicity & Immunogenicity of a 4th Dose of GSK Biologicals' Pneumococcal Vaccine or Prevenar™ in Children (12-18 Months) Previously Vaccinated in the Primary Study NCT00307554 With Either Pneumococcal Vaccine or Prevenar™
Brief Title: Safety and Immunogenicity Study of a Booster Dose of GSK Biologicals' 10-valent Pneumococcal Conjugate Vaccine.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 107046; 2006-001628-38 (EudraCT Number)
Record Dates: First submitted 2006-08-30; First posted 2006-08-31 (Estimated); Results first posted 2018-11-26 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Infections, Streptococcal
Keywords: Streptococcus pneumonia, pneumococcal conjugate vaccine
MeSH Terms: conditions — Streptococcal Infections; Pneumonia | interventions — PHiD-CV vaccine; 10-valent pneumococcal conjugate vaccine; Heptavalent Pneumococcal Conjugate Vaccine; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

ARMS (3):
- Synflorix-Synflorix Group (Experimental): This group consisted of subjects previously vaccinated with the Synflorix™ vaccine as part of a previous study by GSK Biologicals - the 10PN-PD-DIT-001 (105553) study (EuDRA-CT number: 2005-003300-11). As part of the 105553 study, subjects had received a 3-dose primary vaccination of Synflorix™ vaccine at 2, 3 and 4 months of age (injected intramuscularly [IM] in the right thigh) co-administered with Infanrix hexa™ vaccine, except for the second dose in France, which was co-administered with Infanrix™ IPV Hib, injected intramuscularly in the left thigh. As part of this study, at 12-18 months of age, subjects received a booster dose of Synflorix™ vaccine, injected IM in the right thigh or deltoid, co-administered with Infanrix hexa™ vaccine, injected IM in the left thigh or deltoid.
  Interventions: Biological: Synflorix; Biological: Infanrix hexa
- Prevenar-Prevenar Group (Active Comparator): This group consisted of subjects previously vaccinated with the Prevenar™ vaccine as part of a previous study by GSK Biologicals - the 10PN-PD-DIT-001 (105553) study (EuDRA-CT number: 2005-003300-11). As part of the 105553 study, subjects had received a 3-dose primary vaccination of Prevenar™ vaccine at 2, 3 and 4 months of age (injected intramuscularly [IM] in the right thigh) co-administered with Infanrix hexa™ vaccine, except for the second dose in France, which was co-administered with Infanrix™ IPV Hib, injected intramuscularly in the left thigh. As part of this study, at 12-18 months of age, subjects received a booster dose of Prevenar™ vaccine, injected IM in the right thigh or deltoid, co-administered with Infanrix hexa™ vaccine, injected IM in the left thigh or deltoid.
  Interventions: Biological: Prevenar; Biological: Infanrix hexa
- Prevenar-Synflorix Group (Experimental): This group consisted of subjects previously vaccinated with the Prevenar™ vaccine as part of a previous study by GSK Biologicals - the 10PN-PD-DIT-001 (105553) study (EuDRA-CT number: 2005-003300-11). As part of the 105553 study, subjects had received a 3-dose primary vaccination of Synflorix vaccine at 2, 3 and 4 months of age (injected intramuscularly [IM] in the right thigh) co-administered with Infanrix hexa™ vaccine, except for the second dose in France, which was co-administered with Infanrix™ IPV Hib, injected intramuscularly in the left thigh. As part of this study, at 12-18 months of age, subjects received a booster dose of Synflorix™, injected IM in the right thigh or deltoid, co-administered with Infanrix hexa™ vaccine, injected IM in the left thigh or deltoid.
  Interventions: Biological: Synflorix; Biological: Infanrix hexa

INTERVENTIONS:
Biological: Synflorix — 1 dose injected IM in the right thigh or deltoid.
  Other Names: 10 valent pneumococcal conjugate (vaccine)
  Arms: Prevenar-Synflorix Group; Synflorix-Synflorix Group
Biological: Prevenar — 1 dose injected IM in the right thigh or deltoid.
  Arms: Prevenar-Prevenar Group
Biological: Infanrix hexa — 1 dose injected IM in the right thigh or deltoid.

SUMMARY:
This study will evaluate the safety, reactogenicity and immunogenicity of a booster dose of GSK Biologicals' pneumococcal conjugate vaccine compared to Prevenar™ given at 12-18 mo of age to children primed with either pneumococcal vaccine or Prevenar™ in study 105553. Antibody persistence will be evaluated at 8-14 mo after completion of the 3-dose immunization course in study 105553 (NCT00307554). The immune response to a booster dose of GSK Biologicals' pneumococcal conjugate vaccine will also be evaluated when given at 12-18 mo to subjects not primed with GSK Biologicals' vaccine but with Prevenar™.

The study has 3 groups. 1 group of children primed with GSK Biologicals' pneumococcal conjugate vaccine will receive a booster dose of the same vaccine. 2nd group of children primed with Prevenar™ will receive a booster dose of Prevenar™ (control group). 3rd group of children primed with Prevenar™ will receive a booster dose of GSK Biologicals' pneumococcal conjugate vaccine. All children will receive concomitantly a booster dose of DTPa-HBV-IPV/Hib vaccine.

ELIGIBILITY:
Inclusion Criteria:

* a healthy male or female, 12 to 18 months of age at the time of vaccination, who received at least one dose of either pneumococcal conjugate vaccine or Prevenar™ during study 105553 and with written informed consent obtained from the parent/guardian of the subject.

Exclusion Criteria:

* use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding the vaccination, or planned use during the entire study period (active phase and safety follow-up).
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting one month before vaccination up to Visit 2.
* Administration of any additional pneumococcal vaccine or DTPa-combined vaccine since end of study 105553. Children with a history of seizures or neurological disease, allergic disease, immunosuppressive or immunodeficient condition.

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2006-09-25 (Actual); Primary Completion 2007-06-04 (Actual); Study Completion 2007-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (33):
- Finland (14):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Jyväskylä
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Kotka
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vantaa
- France (13):
  - GSK Investigational Site, Bernay
  - GSK Investigational Site, Colombes
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Dax
  - GSK Investigational Site, Draguignan
  - GSK Investigational Site, Essey-lès-Nancy
  - GSK Investigational Site, Le Havre
  - GSK Investigational Site, Maromme
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Nogent-sur-Marne
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Saint-Quentin
- Poland (6):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Oleśnica
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Siemianowice Śląskie

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Wysocki J, Tejedor JC, Grunert D, Konior R, Garcia-Sicilia J, Knuf M, Bernard L, Dieussaert I, Schuerman L. Immunogenicity of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) when coadministered with different neisseria meningitidis serogroup C conjugate vaccines. Pediatr Infect Dis J. 2009 Apr;28(4 Suppl):S77-88. doi: 10.1097/INF.0b013e318199f609. PMID 19325450
- [Background] Chevallier B, Vesikari T, Brzostek J, Knuf M, Bermal N, Aristegui J, Borys D, Cleerbout J, Lommel P, Schuerman L. Safety and reactogenicity of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) when coadministered with routine childhood vaccines. Pediatr Infect Dis J. 2009 Apr;28(4 Suppl):S109-18. doi: 10.1097/INF.0b013e318199f62d. PMID 19325447
- [Background] Knuf M, Szenborn L, Moro M, Petit C, Bermal N, Bernard L, Dieussaert I, Schuerman L. Immunogenicity of routinely used childhood vaccines when coadministered with the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV). Pediatr Infect Dis J. 2009 Apr;28(4 Suppl):S97-S108. doi: 10.1097/INF.0b013e318199f61b. PMID 19325452
- [Background] Silfverdal SA, Coremans V, Francois N, Borys D, Cleerbout J. Safety profile of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV). Expert Rev Vaccines. 2017 Feb;16(2):109-121. doi: 10.1586/14760584.2016.1164044. Epub 2016 Sep 30. PMID 26954689
- [Background] Vesikari T, Wysocki J, Chevallier B, Karvonen A, Czajka H, Arsene JP, Lommel P, Dieussaert I, Schuerman L. Immunogenicity of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) compared to the licensed 7vCRM vaccine. Pediatr Infect Dis J. 2009 Apr;28(4 Suppl):S66-76. doi: 10.1097/INF.0b013e318199f8ef. PMID 19325449
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 107046 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107046 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107046 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107046 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107046 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107046 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of approximately 1200 subjects who were previously enrolled and had been vaccinated with either the 10Pn or 7Pn vaccine as part of the 10PN-PD-DIT-001 (105553) study (EudraCTnumber: 2005-003300-11).
Pre-assignment Details: During the screening the following was performed: informed consent was obtained and signed from parents or guardians of subjects, check for inclusion/exclusion criteria and contraindications/precautions was performed, and medical history of subjects was collected. Prior to vaccination, subjects' pre-vaccination body temperature was evaluated.
Period: Overall Study
Arm/Group | Synflorix-Synflorix Group | Prevenar-Prevenar Group | Prevenar-Synflorix Group
Started (1112 subjects were vaccinated in current study out of 1200 who received at least 1 dose of Prevenar) | 737 | 92 | 283
Completed | 726 | 91 | 282
Not Completed | 11 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lost to Follow-up | 11 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix-Synflorix Group | Prevenar-Prevenar Group | Prevenar-Synflorix Group | Total
Number analyzed (Participants) | 737 | 92 | 283 | 1112
Age, Continuous [Mean (Standard Deviation); unit: Months] | 15.3 (2.08) | 14.2 (2.26) | 14.2 (2.23) | 14.93 (2.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 360 | 50 | 134 | 544
  Male | 377 | 42 | 149 | 568

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Rectal Temperature Above (>) 39.0 Degrees Celsius (°C) Post Booster Between the Synflorix-Synflorix and Prevenar-Prevenar Groups
Description: Fever was measured as rectal temperature. Assessment of occurrences of rectal temperature > 39.0 °C was performed post administration of the booster dose of pneumococcal vaccine (Synflorix™ or Prevenar™ vaccine) in this study. The analysis was performed on the Total vaccinated cohort, which included all subjects vaccinated in this study 10PN-PD-DIT-007, solely on subjects with results available.
Time Frame: Within 4 days (Days 0-3) after the booster vaccination at Month 0 in this study 10PN-PD-DIT-007
Population: The analysis was performed on the Total vaccinated cohort, which included all vaccinated subjects, who completed their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix-Synflorix Group | Prevenar-Prevenar Group
Number analyzed (Participants) | 735 | 91
Participants | 24 | 7
Statistical Analysis 1: Comparison: Synflorix-Synflorix Group vs Prevenar-Prevenar Group; Analysis aimed at demonstrating the non-inferiority of Synflorix™ vs Prevenar™ vaccine, both co-administered with Infanrix hexa™ vaccine, in terms of post-immunization febrile reactions with rectal fever > 39.0°C; Test type: Non-Inferiority or Equivalence — Standardized asymptotic 95% confidence interval (CI) for the difference [Synflorix-Synflorix minus Prevenar-Prevenar] in terms of percentages of subjects reporting rectal fever >39.0°C was computed; Difference in percentage = -4.43, 95% CI 2-sided [-11.85 to -0.21]

2. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling. Grade 3 pain was defined as crying when limb was moved/spontaneously painful. Grade 3 swelling/redness was defined as swelling/redness larger than (>) 30 millimeters (mm). "Any" is defined as incidence of the specified symptom regardless of intensity. The analysis was performed on the Total vaccinated cohort, which included all subjects vaccinated in this study 10PN-PD-DIT-007, solely on subjects with results available.
Time Frame: Within 4 days (Days 0-3) after the booster vaccination at Month 0 in this study 10PN-PD-DIT-007
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix-Synflorix Group | Prevenar-Prevenar Group | Prevenar-Synflorix Group
Number analyzed (Participants) | 735 | 91 | 282
Participants
  Any Pain | 452 | 48 | 150
  Grade 3 Pain | 47 | 3 | 18
  Any Swelling | 338 | 42 | 112
  Grade 3 Swelling | 67 | 7 | 20
  Any Redness | 451 | 59 | 153
  Grade 3 Redness | 96 | 7 | 19

3. Secondary Outcome: Number of Subjects With Any and Any Grade 3 Solicited General Symptoms
Description: Solicited general symptoms assessed include drowsiness, fever (defined as rectal temperature ≥ 38.0°C), irritability, and loss of appetite. Grade 3 drowsiness was defined as drowsiness which prevented normal everyday activities. Grade 3 fever was defined as fever (rectal temperature) above (>) 40.0 degree Celsius (°C). Grade 3 irritability was defined as crying that could not be comforted/preventing normal everyday activities. Grade 3 loss of appetite was defined as the subject not eating at all. "Any" is defined as incidence of the specified symptom regardless of intensity or relationship to study vaccination. The analysis was performed on the Total vaccinated cohort, which included all subjects vaccinated in this study 10PN-PD-DIT-007, solely on subjects with results available.
Time Frame: Within 4 days (Days 0-3) after the booster vaccination at Month 0 in this study 10PN-PD-DIT-007
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix-Synflorix Group | Prevenar-Prevenar Group | Prevenar-Synflorix Group
Number analyzed (Participants) | 735 | 91 | 282
Participants
  Any drowsiness | 303 | 48 | 130
  Grade 3 drowsiness | 5 | 0 | 5
  Any fever | 245 | 33 | 112
  Grade 3 fever | 1 | 2 | 3
  Any irritability | 438 | 55 | 176
  Grade 3 irritability | 15 | 2 | 12
  Any loss of appetite | 230 | 31 | 92
  Grade 3 loss of appetite | 4 | 0 | 3

4. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. "Any" is defined an incidence of an unsolicited AE regardless of intensity or relationship to study vaccination. The analysis was performed on the Total vaccinated cohort, which included all subjects vaccinated in this study 10PN-PD-DIT-007.
Time Frame: Within 31 days (Day 0-30) after the booster vaccination at Month 0 in this study 10PN-PD-DIT-007
Population: The analysis was performed on the Total vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix-Synflorix Group | Prevenar-Prevenar Group | Prevenar-Synflorix Group
Number analyzed (Participants) | 737 | 92 | 283
Participants | 188 | 32 | 99

5. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) During the Active Phase of the Study
Description: An SAE is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or may evolve into one of the outcomes listed above. "Any" is defined an incidence of a SAE regardless of intensity/severity . The analysis was performed on the Total vaccinated cohort, which included all subjects vaccinated in this study 10PN-PD-DIT-007.
Time Frame: Throughout the Active Phase of the study, that is, within 31 days (Day 0-30) after the booster vaccination at Month 0 in this study 10PN-PD-DIT-007
Population: The analysis was performed on the Total vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix-Synflorix Group | Prevenar-Prevenar Group | Prevenar-Synflorix Group
Number analyzed (Participants) | 737 | 92 | 283
Participants | 12 | 1 | 4

6. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) During the Entire Study
Description: An SAE is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or may evolve into one of the outcomes listed above. "Any" is defined an incidence of a SAE regardless of intensity/severity. The analysis was performed on the Total vaccinated cohort, which included all subjects vaccinated in this study 10PN-PD-DIT-007, solely on subjects enrolled in the ESFU Phase of the study.
Time Frame: Throughout the study period, from Month 0 prior to booster vaccination up to Month 6, end of the ESFU in this study 10PN-PD-DIT-007
Population: The analysis was performed on the Total vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix-Synflorix Group | Prevenar-Prevenar Group | Prevenar-Synflorix Group
Number analyzed (Participants) | 726 | 92 | 282
Participants | 33 | 6 | 8

7. Secondary Outcome: Number of Subjects Seroprotected as Regards Anti-pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F Antigens - by 22F-inhibition Enzyme-linked Immunosorbent Assay (ELISA)
Description: A seroprotected subject as regards anti-pneumococcal serotype antibody was defined as a subject with anti-pneumococcal serotype antibody concentration above than or equal to (≥) 0.20 microgram per millilitre (μg/mL). Anti-pneumococcal serotypes antibodies assessed were antibodies against pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Anti-1, -4, -5, -6B, -7F, 9V, -14, -18C, -19F and -23F). Analysis was performed using the 22F-inhibition Enzyme-linked immunosorbent assay (ELISA), using ≥ 0.05 μg/mL as seropositivity cut off. For this endpoint, the analysis was performed on the according-to-protocol cohort for immunogenicity, e. a., evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after booster vaccination.
Time Frame: Prior to (PRE) and one month after (Month 1) booster vaccination
Population: The analysis was performed on the According-To-Protocol (ATP) Cohort for immunogenecity, which included all evaluable subjects whith available immunogenecity data. This included subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after booster vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix-Synflorix Group | Prevenar-Prevenar Group | Prevenar-Synflorix Group
Number analyzed (Participants) | 347 | 89 | 134
Participants
  Anti-1 PRE: number analyzed (Participants) | 338 | 82 | 133
  Anti-1 PRE | 123 | 3 | 3
  Anti-1 Month 1: number analyzed (Participants) | 342 | 81 | 133
  Anti-1 Month 1 | 340 | 4 | 113
  Anti-4 PRE: number analyzed (Participants) | 342 | 78 | 131
  Anti-4 PRE | 196 | 53 | 99
  Anti-4 Month 1: number analyzed (Participants) | 343 | 88 | 133
  Anti-4 Month 1 | 342 | 88 | 133
  Anti-5 PRE: number analyzed (Participants) | 344 | 84 | 134
  Anti-5 PRE | 231 | 5 | 14
  Anti-5 Month 1: number analyzed (Participants) | 342 | 82 | 133
  Anti-5 Month 1 | 340 | 5 | 114
  Anti-6B PRE: number analyzed (Participants) | 333 | 75 | 131
  Anti-6B PRE | 223 | 23 | 69
  Anti-6B Month 1: number analyzed (Participants) | 341 | 87 | 133
  Anti-6B Month 1 | 329 | 85 | 131
  Anti-7F PRE: number analyzed (Participants) | 340 | 85 | 133
  Anti-7F PRE | 308 | 4 | 3
  Anti-7F Month 1: number analyzed (Participants) | 342 | 85 | 133
  Anti-7F Month 1 | 342 | 6 | 127
  Anti-9V PRE: number analyzed (Participants) | 344 | 77 | 130
  Anti-9V PRE | 291 | 70 | 123
  Anti-9V Month 1: number analyzed (Participants) | 340 | 89 | 133
  Anti-9V Month 1 | 340 | 89 | 133
  Anti-14 PRE: number analyzed (Participants) | 336 | 75 | 130
  Anti-14 PRE | 268 | 70 | 125
  Anti-14 Month 1: number analyzed (Participants) | 339 | 86 | 133
  Anti-14 Month 1 | 336 | 86 | 133
  Anti-18C PRE: number analyzed (Participants) | 341 | 83 | 131
  Anti-18C PRE | 240 | 60 | 107
  Anti-18C Month 1: number analyzed (Participants) | 343 | 87 | 134
  Anti-18C Month 1 | 343 | 87 | 133
  Anti-19F PRE: number analyzed (Participants) | 347 | 85 | 134
  Anti-19F PRE | 272 | 38 | 76
  Anti-19F Month 1: number analyzed (Participants) | 343 | 87 | 134
  Anti-19F Month 1 | 341 | 87 | 131
  Anti-23F PRE: number analyzed (Participants) | 338 | 77 | 130
  Anti-23F PRE | 206 | 43 | 98
  Anti-23F Month 1: number analyzed (Participants) | 341 | 88 | 132
  Anti-23F Month 1 | 332 | 87 | 128

8. Secondary Outcome: Antibody Concentrations Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Anti-1, -4, -5, -6B, -7F, 9V, -14, -18C, -19F and -23F) - by 22F-inhibition Enzyme-linked Immunosorbent Assay (ELISA)
Description: Anti-pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F antibody concentrations (Anti-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F) were calculated, expressed as geometric mean concentrations (GMCs), in microgram per millilitre (µg/mL). The seropositivity cut-off for the assay was ≥ 0.05 µg/mL. Antibody concentrations below the cut-off of the assay were given an arbitrary value of half the cut-off for the purpose of GMC calculation. For this endpoint, the analysis was performed on the according-to-protocol cohort for immunogenicity, e. a., evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after booster vaccination.
Time Frame: Prior to (PRE) and one month (Month 1) post booster vaccination
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix-Synflorix Group | Prevenar-Prevenar Group | Prevenar-Synflorix Group
Number analyzed (Participants) | 347 | 89 | 134
μg/mL
  Anti-1 PRE: number analyzed (Participants) | 338 | 82 | 133
  Anti-1 PRE | 0.14 [0.13 to 0.16] | 0.03 [0.03 to 0.04] | 0.03 [0.03 to 0.04]
  Anti-1 Month 1: number analyzed (Participants) | 342 | 81 | 133
  Anti-1 Month 1 | 1.53 [1.4 to 1.68] | 0.04 [0.03 to 0.05] | 0.67 [0.56 to 0.8]
  Anti-4 PRE: number analyzed (Participants) | 342 | 78 | 131
  Anti-4 PRE | 0.23 [0.21 to 0.26] | 0.3 [0.25 to 0.37] | 0.35 [0.3 to 0.41]
  Anti-4 Month 1: number analyzed (Participants) | 343 | 88 | 133
  Anti-4 Month 1 | 3.35 [3.06 to 3.67] | 4.4 [3.75 to 5.15] | 4.47 [3.85 to 5.19]
  Anti-5 PRE: number analyzed (Participants) | 344 | 84 | 134
  Anti-5 PRE | 0.27 [0.25 to 0.3] | 0.04 [0.04 to 0.05] | 0.05 [0.04 to 0.05]
  Anti-5 Month 1: number analyzed (Participants) | 342 | 82 | 133
  Anti-5 Month 1 | 2.2 [2 to 2.42] | 0.05 [0.04 to 0.07] | 0.74 [0.6 to 0.9]
  Anti-6B PRE: number analyzed (Participants) | 333 | 75 | 131
  Anti-6B PRE | 0.31 [0.27 to 0.35] | 0.14 [0.11 to 0.19] | 0.26 [0.2 to 0.33]
  Anti-6B Month 1: number analyzed (Participants) | 341 | 87 | 133
  Anti-6B Month 1 | 1.94 [1.74 to 2.17] | 3.53 [2.83 to 4.41] | 1.74 [1.48 to 2.05]
  Anti-7F PRE: number analyzed (Participants) | 340 | 85 | 133
  Anti-7F PRE | 0.57 [0.52 to 0.62] | 0.03 [0.03 to 0.04] | 0.03 [0.03 to 0.03]
  Anti-7F Month 1: number analyzed (Participants) | 342 | 85 | 133
  Anti-7F Month 1 | 3.5 [3.25 to 3.76] | 0.04 [0.03 to 0.05] | 1.83 [1.49 to 2.24]
  Anti-9V PRE: number analyzed (Participants) | 344 | 77 | 130
  Anti-9V PRE | 0.54 [0.48 to 0.6] | 0.62 [0.51 to 0.76] | 0.78 [0.68 to 0.89]
  Anti-9V Month 1: number analyzed (Participants) | 340 | 89 | 133
  Anti-9V Month 1 | 3.25 [2.99 to 3.53] | 6.09 [5.19 to 7.15] | 1.94 [1.73 to 2.19]
  Anti-14 PRE: number analyzed (Participants) | 336 | 75 | 130
  Anti-14 PRE | 0.66 [0.56 to 0.76] | 1.06 [0.82 to 1.38] | 1.69 [1.4 to 2.03]
  Anti-14 Month 1: number analyzed (Participants) | 339 | 86 | 133
  Anti-14 Month 1 | 5.56 [5.01 to 6.18] | 9.29 [7.85 to 10.99] | 4.76 [4.12 to 5.49]
  Anti-18C PRE: number analyzed (Participants) | 341 | 83 | 131
  Anti-18C PRE | 0.3 [0.28 to 0.34] | 0.32 [0.26 to 0.39] | 0.37 [0.32 to 0.43]
  Anti-18C Month 1: number analyzed (Participants) | 343 | 87 | 134
  Anti-18C Month 1 | 5.01 [4.6 to 5.46] | 5.21 [4.44 to 6.11] | 4.98 [4.17 to 5.93]
  Anti-19F PRE: number analyzed (Participants) | 347 | 85 | 134
  Anti-19F PRE | 0.53 [0.46 to 0.61] | 0.23 [0.17 to 0.31] | 0.31 [0.24 to 0.41]
  Anti-19F Month 1: number analyzed (Participants) | 343 | 87 | 134
  Anti-19F Month 1 | 6.05 [5.46 to 6.71] | 3.35 [2.83 to 3.97] | 5.06 [4.24 to 6.04]
  Anti-23F PRE: number analyzed (Participants) | 338 | 77 | 130
  Anti-23F PRE | 0.27 [0.23 to 0.31] | 0.24 [0.19 to 0.31] | 0.4 [0.3 to 0.5]
  Anti-23F Month 1: number analyzed (Participants) | 341 | 88 | 132
  Anti-23F Month 1 | 2.38 [2.13 to 2.66] | 6.67 [5.38 to 8.26] | 2.42 [1.99 to 2.95]

9. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F
Description: OPA titers against pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Opsono-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F) were calculated, expressed as geometric mean titers (GMTs) and tabulated. The seropositivity cut-off for the assay was ≥ 8. Antibody titers below the cut-off of the assay were given an arbitrary value of half the cut-off for the purpose of GMT calculation. For this endpoint, the analysis was performed on the according-to-protocol cohort for immunogenicity, e. a., evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after booster vaccination.
Time Frame: Prior to (PRE) and one month (Month 1) post booster vaccination
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix-Synflorix Group | Prevenar-Prevenar Group | Prevenar-Synflorix Group
Number analyzed (Participants) | 326 | 83 | 126
Titers
  Opsono-1 PRE | 6.1 [5.4 to 6.9] | 5 [4.1 to 6] | 4.9 [4.2 to 5.8]
  Opsono-1 Month 1: number analyzed (Participants) | 301 | 83 | 121
  Opsono-1 Month 1 | 192.2 [157.5 to 234.6] | 4.3 [3.9 to 4.7] | 8.3 [6.7 to 10.4]
  Opsono-4 PRE: number analyzed (Participants) | 295 | 79 | 112
  Opsono-4 PRE | 20.3 [16.2 to 25.5] | 24.5 [15.4 to 38.8] | 37.8 [24.8 to 57.7]
  Opsono-4 Month 1: number analyzed (Participants) | 297 | 81 | 123
  Opsono-4 Month 1 | 1856.3 [1666.1 to 2068] | 2812.6 [2282.5 to 3465.9] | 1528.9 [1286.9 to 1817]
  Opsono-5 PRE: number analyzed (Participants) | 305 | 79 | 124
  Opsono-5 PRE | 8.2 [7.2 to 9.4] | 4.4 [3.9 to 4.9] | 4.1 [3.9 to 4.3]
  Opsono-5 Month 1: number analyzed (Participants) | 299 | 83 | 122
  Opsono-5 Month 1 | 144.1 [122.1 to 170] | 4.1 [3.9 to 4.4] | 9.5 [7.5 to 11.9]
  Opsono-6B PRE: number analyzed (Participants) | 284 | 75 | 120
  Opsono-6B PRE | 60.3 [44.6 to 81.7] | 51.4 [27.1 to 97.5] | 36.7 [23.3 to 57.7]
  Opsono-6B Month 1: number analyzed (Participants) | 295 | 79 | 118
  Opsono-6B Month 1 | 981.2 [830.7 to 1159.1] | 3459.6 [2535.7 to 4720.3] | 640.2 [480.7 to 852.7]
  Opsono-7F PRE: number analyzed (Participants) | 294 | 76 | 117
  Opsono-7F PRE | 377.7 [279.8 to 509.9] | 34.8 [17.5 to 69.3] | 25.3 [15.4 to 41.6]
  Opsono-7F Month 1: number analyzed (Participants) | 296 | 74 | 118
  Opsono-7F Month 1 | 4330.3 [3836 to 4888.3] | 25.2 [13.1 to 48.7] | 2397.2 [1929.2 to 2978.7]
  Opsono-9V PRE: number analyzed (Participants) | 309 | 81 | 122
  Opsono-9V PRE | 296.9 [259.3 to 339.9] | 305.5 [227.1 to 411] | 305.1 [248.7 to 374.4]
  Opsono-9V Month 1: number analyzed (Participants) | 297 | 79 | 120
  Opsono-9V Month 1 | 2343.5 [2097.1 to 2618.7] | 5357.4 [4212.5 to 6813.6] | 886.8 [747.7 to 1051.8]
  Opsono-14 PRE: number analyzed (Participants) | 299 | 79 | 118
  Opsono-14 PRE | 188.1 [149.9 to 235.9] | 201.6 [129.4 to 314.2] | 391.1 [303.1 to 504.6]
  Opsono-14 Month 1: number analyzed (Participants) | 304 | 82 | 123
  Opsono-14 Month 1 | 2085.9 [1868 to 2329.1] | 2134.2 [1689.1 to 2696.6] | 977.8 [828.9 to 1153.5]
  Opsono-18C PRE: number analyzed (Participants) | 309 | 82 | 121
  Opsono-18C PRE | 8.7 [7.4 to 10.3] | 10.4 [7.4 to 14.7] | 8.5 [6.6 to 10.9]
  Opsono-18C Month 1: number analyzed (Participants) | 299 | 76 | 121
  Opsono-18C Month 1 | 810.3 [712.4 to 921.7] | 968.7 [724.1 to 1295.8] | 610.7 [480.3 to 776.4]
  Opsono-19F PRE: number analyzed (Participants) | 317 | 81 | 123
  Opsono-19F PRE | 10.5 [8.9 to 12.3] | 5.9 [4.5 to 7.8] | 7.3 [5.5 to 9.6]
  Opsono-19F Month 1: number analyzed (Participants) | 293 | 80 | 120
  Opsono-19F Month 1 | 624.3 [509.7 to 764.7] | 287.8 [190.8 to 434.3] | 530.1 [393 to 715.2]
  Opsono-23F PRE: number analyzed (Participants) | 305 | 77 | 120
  Opsono-23F PRE | 171.5 [126.3 to 232.8] | 205.8 [110.1 to 384.6] | 532.9 [344.4 to 824.7]
  Opsono-23F Month 1: number analyzed (Participants) | 301 | 80 | 121
  Opsono-23F Month 1 | 2830.1 [2487.2 to 3220.3] | 13900.7 [10177.4 to 18986.1] | 2828.8 [2234.3 to 3581.6]

10. Secondary Outcome: Antibody Concentrations to Protein D (Anti-PD) - by Enzyme-Linked Immunosorbent Assay (ELISA)
Description: Anti-protein D (Anti-PD) antibody concentrations by Enzyme-Linked Immunosorbent Assay (ELISA) were calculated, expressed as geometric mean concentrations (GMCs) in ELISA unit per milli-liter (EL.U/mL) and tabulated. The seropositivity cut-off for the assay was ≥ 100 EL.U/mL. Antibody concentrations below the cut-off of the assay were given an arbitrary value of half the cut-off for the purpose of GMC calculation. For this endpoint, the analysis was performed on the according-to-protocol cohort for immunogenicity, e. a., evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after booster vaccination.
Time Frame: Prior to (PRE) and one month (Month 1) post booster vaccination
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix-Synflorix Group | Prevenar-Prevenar Group | Prevenar-Synflorix Group
Number analyzed (Participants) | 340 | 86 | 134
EL.U/mL
  Anti-PD, PRE: number analyzed (Participants) | 338 | 73 | 127
  Anti-PD, PRE | 556.4 [494.7 to 625.7] | 72.3 [59.3 to 88] | 78.1 [67.8 to 89.9]
  Anti-PD, Month 1 | 2887.6 [2573.7 to 3239.8] | 75.3 [60 to 94.4] | 125.5 [103.4 to 152.4]

11. Secondary Outcome: Anti-polyribosyl Ribitol Phosphate (Anti-PRP) Antibody Concentrations
Description: Anti-PRP antibody concentrations were calculated, expressed as geometric mean concentrations (GMCs), in microgram per milliliter (µg/mL), and tabulated. The seroprotection cut-off for the assay for the purpose of this endpoint was ≥ 0.15 µg/mL. Antibody concentrations below the cut-off of the assay were given an arbitrary value of half the cut-off for the purpose of GMC calculation. For this endpoint, the analysis was performed on the according-to-protocol cohort for immunogenicity, e. a., evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after booster vaccination.
Time Frame: Prior to (PRE) and one month (Month 1) post booster vaccination
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix-Synflorix Group | Prevenar-Prevenar Group | Prevenar-Synflorix Group
Number analyzed (Participants) | 344 | 46 | 136
μg/mL
  Anti-PRP, PRE: number analyzed (Participants) | 344 | 39 | 136
  Anti-PRP, PRE | 0.308 [0.272 to 0.348] | 0.231 [0.151 to 0.353] | 0.246 [0.2 to 0.304]
  Anti-PRP, Month 1: number analyzed (Participants) | 343 | 46 | 136
  Anti-PRP, Month 1 | 36.634 [31.897 to 42.074] | 25.731 [15.87 to 41.719] | 29.851 [23.563 to 37.816]

12. Secondary Outcome: Anti-pertussis Toxoid (Anti-PT), Anti- Filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibody Concentrations
Description: Anti-PT, Anti-FHA and Anti-PRN concentrations measured by Enzyme-Linked Immunosorbent Assay (ELISA) were calculated, expressed as geometric mean concentrations (GMCs) in ELISA unit per milli-liter (EL.U/mL) and tabulated. The seropositivity cut-off for the assay was ≥ 5 EL.U/mL. Antibody concentrations below the cut-off of the assay were given an arbitrary value of half the cut-off for the purpose of GMC calculation. For this endpoint, the analysis was performed on the according-to-protocol cohort for immunogenicity, e. a., evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after booster vaccination.
Time Frame: Prior to (PRE) and one month (Month 1) post booster vaccination
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix-Synflorix Group | Prevenar-Prevenar Group | Prevenar-Synflorix Group
Number analyzed (Participants) | 344 | 46 | 136
EL.U/mL
  Anti-PT, PRE: number analyzed (Participants) | 332 | 34 | 133
  Anti-PT, PRE | 5.5 [5.1 to 6.1] | 7.3 [5.2 to 10.3] | 7 [6.1 to 8.1]
  Anti-PT, Month 1: number analyzed (Participants) | 338 | 46 | 135
  Anti-PT, Month 1 | 79.6 [73.8 to 85.9] | 76 [60.4 to 95.7] | 85.8 [76.9 to 95.7]
  Anti-FHA, PRE: number analyzed (Participants) | 343 | 36 | 135
  Anti-FHA, PRE | 27.1 [24.4 to 30.1] | 29 [20.5 to 40.8] | 35.5 [29.7 to 42.3]
  Anti-FHA, Month 1: number analyzed (Participants) | 343 | 46 | 136
  Anti-FHA, Month 1 | 357.7 [332.6 to 384.7] | 334.5 [278.1 to 402.2] | 400.2 [356.4 to 449.5]
  Anti-PRN, PRE: number analyzed (Participants) | 344 | 34 | 136
  Anti-PRN, PRE | 9.1 [8.2 to 10.1] | 11.1 [7.6 to 16.2] | 12.1 [10.1 to 14.6]
  Anti-PRN, Month 1: number analyzed (Participants) | 342 | 45 | 135
  Anti-PRN, Month 1 | 248.9 [226.5 to 273.4] | 204.6 [155.8 to 268.7] | 276.5 [239.1 to 319.7]

13. Secondary Outcome: Anti-diphtheria (Anti-D) and Anti-tetanus Toxoids (Anti-TT) Antibody Concentrations
Description: Anti-D and Anti-TT antibody concentrations were calculated, expressed as geometric mean concentrations (GMCs), in International units per milliliter (IU/mL), and tabulated. The seropositivity cut-off for the assay was ≥ 0.1 IU/mL. Antibody concentrations below the cut-off of the assay were given an arbitrary value of half the cut-off for the purpose of GMC calculation. For this endpoint, the analysis was performed on the according-to-protocol cohort for immunogenicity, e. a., evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after booster vaccination.
Time Frame: Prior to (PRE) and one month (Month 1) post booster vaccination
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix-Synflorix Group | Prevenar-Prevenar Group | Prevenar-Synflorix Group
Number analyzed (Participants) | 344 | 46 | 136
EL.U/mL
  Anti-D, PRE: number analyzed (Participants) | 344 | 34 | 136
  Anti-D, PRE | 0.179 [0.161 to 0.199] | 0.291 [0.2 to 0.424] | 0.29 [0.25 to 0.336]
  Anti-D, Month 1: number analyzed (Participants) | 343 | 45 | 136
  Anti-D, Month 1 | 5.809 [5.352 to 6.305] | 6.272 [4.883 to 8.055] | 9.337 [8.419 to 10.356]
  Anti-TT, PRE: number analyzed (Participants) | 344 | 35 | 136
  Anti-TT, PRE | 0.417 [0.382 to 0.456] | 0.261 [0.187 to 0.364] | 0.265 [0.225 to 0.313]
  Anti-TT, Month 1: number analyzed (Participants) | 343 | 46 | 136
  Anti-TT, Month 1 | 9.983 [9.293 to 10.724] | 4.28 [3.294 to 5.562] | 5.677 [5.038 to 6.397]

14. Secondary Outcome: Anti-hepatitis B Surface Antigen (HBs) Antibody Concentrations
Description: Anti-HBs antibody concentrations were calculated, expressed as geometric mean concentrations (GMCs), in milli-International unit per milliliter (IU/mL), and tabulated. The seropositivity cut-off for the assay was ≥ 10 mIU/mL. Antibody concentrations below the cut-off of the assay were given an arbitrary value of half the cut-off for the purpose of GMC calculation. For this endpoint, the analysis was performed on the according-to-protocol cohort for immunogenicity, e. a., evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after booster vaccination.
Time Frame: Prior to (PRE) and one month (Month 1) post booster vaccination
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Synflorix-Synflorix Group | Prevenar-Prevenar Group | Prevenar-Synflorix Group
Number analyzed (Participants) | 329 | 48 | 134
mIU/mL
  Anti-HBs, PRE | 147.2 [124.7 to 173.7] | 148.9 [100.4 to 220.8] | 156.6 [125.5 to 195.5]
  Anti-HBs, Month 1: number analyzed (Participants) | 325 | 47 | 132
  Anti-HBs, Month 1 | 3869.1 [3218.1 to 4651.8] | 3132.2 [1906.3 to 5146.5] | 4358.6 [3495.5 to 5434.8]

15. Secondary Outcome: Anti-polio Type 1, 2 and 3 (Anti-Polio 1, 2 and 3) Antibody Titers
Description: Anti-Polio 1, 2 and 3 antibody titers were calculated, expressed as geometric mean titers (GMTs) and tabulated. The seroprotection cut-off for the assay was ≥ 8. Antibody titers below the cut-off of the assay were given an arbitrary value of half the cut-off for the purpose of GMT calculation. For this endpoint, the analysis was performed on the according-to-protocol cohort for immunogenicity, e. a., evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after booster vaccination.
Time Frame: Prior to (PRE) and one month (Month 1) post booster vaccination
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix-Synflorix Group | Prevenar-Prevenar Group | Prevenar-Synflorix Group
Number analyzed (Participants) | 318 | 48 | 131
Titers
  Anti-Polio 1, PRE | 25.3 [21.9 to 29.3] | 21.2 [15 to 30] | 27.1 [20.7 to 35.4]
  Anti-Polio 1, Month 1: number analyzed (Participants) | 279 | 42 | 121
  Anti-Polio 1, Month 1 | 904.4 [779.7 to 1049.1] | 819.3 [552.9 to 1214.2] | 1003.7 [817.5 to 1232.3]
  Anti-Polio 2, PRE: number analyzed (Participants) | 317 | 46 | 130
  Anti-Polio 2, PRE | 20.8 [18.1 to 24] | 12.9 [8.8 to 18.9] | 17.9 [14.1 to 22.8]
  Anti-Polio 2 , Month 1 | 793.5 [679.7 to 926.3] | 495.7 [300.2 to 818.5] | 661.2 [496.7 to 880.3]
  Anti-Polio 3, PRE: number analyzed (Participants) | 262 | 39 | 113
  Anti-Polio 3, PRE | 33.7 [28.5 to 39.8] | 25.8 [16.7 to 39.8] | 28.2 [21.6 to 36.8]
  Anti-Polio 3, Month 1: number analyzed (Participants) | 270 | 41 | 116
  Anti-Polio 3, Month 1 | 1465 [1257.1 to 1707.3] | 1191.7 [743.1 to 1911.3] | 1646.5 [1294.4 to 2094.5]

16. Secondary Outcome: Number of Subjects Booster (BST) Responder to Pertussis Toxoid (PT), Filamentous Haemagglutinin (FHA) and Pertactin Antigens
Description: A BST responder to PT, FHA and PRN antigens was defined as a subject with the appearance of antibodies in subjects who were seronegative prior to the booster vaccination or at least 2-fold increase of pre-booster vaccination antibody concentrations in subjects who were seropositive prior to the booster vaccination. A seropositive/seronegative subject as regards Anti-PT/-FHA/ -PRN antibodies was defined as a subject with anti-PT/-FHA/ -PRN antibody concentrations ≥ 5 Enzyme-linked Immunosorbent assay (ELISA) unit per milli-liter (EL.U/mL)
Time Frame: One month (Month 1) post booster vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix-Synflorix Group | Prevenar-Prevenar Group | Prevenar-Synflorix Group
Number analyzed (Participants) | 340 | 33 | 135
Participants
  BST responder to PT antigens: number analyzed (Participants) | 324 | 31 | 132
  BST responder to PT antigens | 323 | 31 | 132
  BST responder to FHA antigens | 332 | 31 | 129
  BST responder to PRN antigens: number analyzed (Participants) | 340 | 31 | 135
  BST responder to PRN antigens | 339 | 30 | 131

ADVERSE EVENTS:
Time Frame: From Month 1 (Active Phase) and up to Month 6 (Extended Safety Follow-Up)
Arm/Group | Synflorix-Synflorix Group | Prevenar-Prevenar Group | Prevenar-Synflorix Group
All-Cause Mortality (participants affected / at risk) | 0/737 | 0/92 | 0/283
Serious Adverse Events (participants affected / at risk) | 33/737 | 6/92 | 8/93
Other Adverse Events (participants affected / at risk) | 684/737 | 85/92 | 253/283
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Synflorix-Synflorix Group (N=737) | Prevenar-Prevenar Group (N=92) | Prevenar-Synflorix Group (N=93)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (3) | 1 (1) | 4 (4)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 9 (9) | 0 (0) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Weight gain poor (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 2 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Synflorix-Synflorix Group (N=737) | Prevenar-Prevenar Group (N=92) | Prevenar-Synflorix Group (N=283)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3) | 14 (14)
Decreased appetite (Metabolism and nutrition disorders) | 230 (230) | 31 (31) | 92 (92)
Erythema (Skin and subcutaneous tissue disorders) | 454 (454) | 59 (59) | 153 (154)
Injection site induration (General disorders) | 1 (1) | 7 (7) | 7 (7)
Irritability (Psychiatric disorders) | 438 (438) | 55 (56) | 176 (179)
Otitis media (Infections and infestations) | 16 (17) | 4 (6) | 11 (12)
Pain (General disorders) | 452 (452) | 48 (48) | 150 (150)
Pyrexia (General disorders) | 254 (254) | 35 (36) | 118 (124)
Rhinitis (Infections and infestations) | 28 (28) | 4 (5) | 19 (20)
Somnolence (Nervous system disorders) | 303 (303) | 48 (48) | 130 (130)
Swelling (General disorders) | 338 (339) | 42 (42) | 139 (139)
Upper respiratory tract infection (Infections and infestations) | 24 (24) | 5 (6) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.